CLINICAL TRIAL: NCT04394559
Title: Prevention of Opioid Use Disorder After Surgery: A Pilot and Feasibility Study
Brief Title: Prevention of Opioid Use Disorder After Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Principal Investigator, Jeffrey L. Schnipper, MD.,MPH., Medical Doctor, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020P001387
Record Dates: First submitted 2020-05-10; First posted 2020-05-19 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Opioid-use Disorder; Opioid Dependence; Opioid Use
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Other: 2 arms, before-after study and mixed methods analysis of implementation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): inpatient pharmacists as available; standard discharge orders; standard follow up visit.
- Intervention (Experimental): Discharge counseling; discharge opioid order set; post-discharge pain management follow up; patient pain management app.
  Interventions: Behavioral: Discharge Order Sets; Behavioral: Pharmacist-Led Discharge Counseling and Communication; Behavioral: Post-discharge Pain Management Follow-up; Behavioral: Patient Engagement Pain Management App

INTERVENTIONS:
Behavioral: Discharge Order Sets — Discharge order sets will be implemented in the electronic health record and will provide surgeons a guideline for a recommended dose and duration of opioids for each commonly performed orthopedic surgery.
  Arms: Intervention
Behavioral: Pharmacist-Led Discharge Counseling and Communication — Two visits by a trained inpatient pharmacist, including an intake visit to determine previous barriers to safe medication use, and a discharge counseling session with patients and caregivers regarding safe and effective opioid use after discharge; pharmacist communication with providers regarding the post-discharge pain management plan.
  Arms: Intervention
Behavioral: Post-discharge Pain Management Follow-up — An outpatient pharmacist pain management follow-up visit (with additional contact as needed) embedded within routine post-operative care for managing pain and opioid use.
  Arms: Intervention
Behavioral: Patient Engagement Pain Management App — A mobile patient-reported outcomes application for assessing pain, function, and possible development of opioid use disorder.
  Arms: Intervention

SUMMARY:
The objective of this study is to design, implement, and pilot test a multi-faceted intervention to support safer opioid prescribing, self-administration, and monitoring and reduce persistent opioid use and opioid use disorder for patients transitioning to the community setting after major orthopedic surgery. The multi-faceted intervention includes: 1) communication with outpatient providers and counseling of patients and caregivers at hospital discharge; 2) standardized opioid prescribing discharge order sets for each type of surgery; 3) an outpatient pain management follow-up visit embedded within routine post-operative care for managing pain and opioid use, and 4) a mobile patient-reported outcomes application for assessing pain, function, and possible development of opioid use disorder (OUD). The primary outcome will be persistent opioid use (in the 6 months after surgery) based on state-wide prescription data. Secondary outcomes will include the total morphine-equivalent dose of opioids prescribed at discharge; total post-operative opioids dispensed in the 6 months after surgery; and self-reported opioid misuse, pain and function 90 and 180 days after surgery.

DETAILED DESCRIPTION:
In this study, we will enroll patients who are both opioid-naïve and non-naïve who have undergone orthopedic surgery. To minimize contamination and best evaluate implementation, we will conduct a before-after study. The intervention will consist of four main components: 1) pharmacist-led discharge counseling and communication, 2) discharge order sets, 3) post-discharge pain management follow-up visits; and 4) a patient engagement pain management app. The intervention will last for 6 months following hospital discharge. We plan to enroll 270 patients over a 6-month period to demonstrate the feasibility of the intervention and provide reasonable precision on an effect size to inform power calculations on a subsequent larger scale clinical trial. During implementation, we will measure intervention fidelity and conduct qualitative interviews of stakeholders regarding facilitators and barriers to implementation. Throughout the study, we will engage a patient-family advisory council, other stakeholders, and a Steering Committee and Working Group to guide development and refinement of the intervention, execution of the implementation and evaluation plan, and the communication plan.

Specific Aims:

* Aim 1: To design and implement a multi-faceted intervention (MOPP) to minimize persistent post-operative opioid use while providing adequate analgesia in patients who are status post major orthopedic surgery.
* Aim 2: To pilot test and evaluate the efficacy of MOPP on preventing persistent postoperative opioid use while maintaining adequate analgesia and functional status.
* Aim 3: To evaluate the feasibility and the success of implementation of MOPP and identify barriers to and facilitators of implementation by using mixed methods and the Consolidated Framework for Implementation Research (CFIR).

In the first 3 months of the study, patients will be assigned to usual care, including 1) multimodal analgesia after surgery; 2) unit-based pharmacists as available to monitor the appropriateness of inpatient medication orders, including opioids; 3) the standard discharge medication reconciliation module in the electronic health record (EHR) that compares preadmission and current inpatient medications to facilitate writing of safe medication orders; 4) general guidelines to limit the dose and duration of discharge opioids and to council patients about tapering opioids at home and to stop them by 4-6 weeks post-operatively unless instructed otherwise; and 5) standard follow-up in the outpatient orthopedics clinic within a time frame judged to be appropriate by each inpatient team. In months 4-6 of the study, patients will be assigned to the intervention. The intervention, which we will refer to as MOPP, will consist of four complementary components, as explained below. Each of these is in addition to usual care, as described above.

1. Pharmacist-Led Discharge Counseling and Communication: Based on previously designed and evaluated interventions, an inpatient pharmacist will visit each intervention patient on two occasions: 1) An initial intake visit to screen for previous barriers to safe medication use, including lack of understanding of medication regimens, non-adherence, previous side effects, prior substance use disorder or current misuse of substances other than opioids, and lack of monitoring; 2) Prior to discharge and after the discharge opioid regimen has been determined, to provide counseling regarding safe medication use after discharge, address any of the barriers identified from the intake visit, and specifically cover several topics related to safe opioid use.
2. Discharge Order Sets: One of the challenges to opioid safety following surgery is the large variation in the dose and duration of opioids prescribed at hospital discharge. Therefore, the first step in developing a discharge order set will be generating consensus among the orthopedic surgeons for a recommended dose and duration of opioids for each commonly performed orthopedic surgery. Following this standardization process, we will work with Partners Information Systems to create a discharge order set for all orthopedic patients. It will include embedded decision support where providers can enter the orthopedic surgery type and receive the recommended discharge opioid regimen. Ordering providers will still be able to prescribe doses, frequencies, and durations other than the recommended amount, but the order set will provide a default.
3. Post-Discharge Pain Management Follow-Up: We've chosen to utilize a clinical pharmacist trained in the principles of safe opioid use and pain management to serve as the outpatient pain management follow-up clinician. Follow-up will take place in the outpatient orthopedics department so that patients can see this follow-up clinician as part of already scheduled visits with the orthopedic surgeon and staff after returning home. During the initial post-discharge visit, the focus will be on pain control, functional status, use of opioids and other analgesics, and screening for any possible misuse of opioids. Based on this information, the pharmacist will work with the patient's orthopedist on an action plan, including changes to the patient's opioid regimen, plans for tapers or discontinuation, etc. If there are concerns for development of OUD, then proper referrals and communication will be made to the outpatient addiction psychiatry service. Finally, additional office visits and/or follow-up phone calls will be scheduled as needed. We will maintain an electronic registry of all the patients in the intervention arm so the outpatient pharmacist can track all patients who may have been lost to follow-up, readmitted to the hospital, or have concerning opioid orders, and intervene as necessary.
4. Patient Engagement Pain Management App: Based on the version already created for patients with chronic opioid use, the app will be designed to collect and communicate patient-reported outcomes regarding pain management after discharge. Using the app, patients will be able to rate their current pain, including its effects on sleep, function, and mood, and whether their pain is improving or getting worse. We also plan to link the app to the patient's currently prescribed analgesic regimen so that patients can quickly record how they are taking their medications (compared with how they are prescribed). Patients will also have the ability to securely communicate with their outpatient pain management pharmacist for concerns or questions. The research staff will check the server daily for 2-way messages and link the data to the electronic medical record. Other modifications, including a Spanish version and changes unique to this post-orthopedic surgery patient population, will be made during the first 9 months of the study period based on user input and pilot testing.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to orthopedic or neuro-surgical spine services at Brigham and Women's Hospital during the 6 month enrollment period
* English or Spanish speakers
* Patients who are and are not opioid-naïve for 30 days prior to admission based on their verified preadmission medication list and state-wide opioid prescription information.
* Undergo one of several designated orthopedic or spine surgeries, including trauma and arthroplasty surgeries.
* Age 18 or older
* Clinical discharge plan to home or short-term rehabilitation facility.

Exclusion Criteria:

* Not pregnant women, prisoners or institutionalized individuals
* Under the age of 18
* Current illicit opioid use.
* Patient is unable to provide informed consent, and has no available proxy
* Plan to be discharged to an acute care facility.
* Patient requires a second surgery or has medical condition requiring opioid use during the 6-month follow-up period (data are censored at time of second surgery).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Persistent Opioid Use | Post intervention: 90 days after discharge
  From prescription monitoring program (PMP) data, at least one filled opioid prescription 0-90 days after discharge and another 91-180 days after discharge.
Persistent Opioid Use | Post intervention: 180 days after discharge
  From prescription monitoring program (PMP) data, at least one filled opioid prescription 0-90 days after discharge and another 91-180 days after discharge.

SECONDARY OUTCOMES:
Long-term Opioid Episodes | 180 days after discharge
  From prescription monitoring program (PMP), 3 or more opioid prescriptions dispensed at least 21 days apart; a duration of at least 84 days between the first day of the first prescription and the last day of the last prescription; and at least 84 days of opioids supplied.
Pain Levels Post-Surgery | 90 days after discharge
  Brief Pain Inventory (BPI), 0-10 scales in 9 categories.
Pain Levels Post-Surgery | 180 days after discharge
  Brief Pain Inventory (BPI), 0-10 scales in 9 categories.
Function | 90 days after discharge
  Patient-Reported Outcomes Measurement Information System- Pain Interference (PROMIS-PI), 0-5 scales.
Function | 180 days after discharge
  Patient-Reported Outcomes Measurement Information System- Pain Interference (PROMIS-PI), 0-5 scales.
Risk of Opioid Use Disorder (OUD) | 90 days after discharge
  Current Opioid Misuse Measure (COMM), 0-4 scales in 17 items.
Risk of Opioid Use Disorder (OUD) | 180 days after discharge
  Current Opioid Misuse Measure (COMM), 0-4 scales in 17 items.
Opioid Use on Discharge | At day 1 at the time of discharge
  From discharge orders, morphine equivalent dose (MED) of the opioids prescribed at discharge using the opioid type, route, dose, maximum frequency, and duration.
Total Post-operative Opioid Use | 180 days after discharge
  From PMP data, total MED of all opioids prescribed and dispensed during the study period.
Post-operative Health Care Utilization | 180 days after discharge
  From health system administrative data (for utilization within Partners Healthcare) plus patient self-report (for utilization outside Partners). Emergency Department visits and hospital admissions, measured as any health care utilization and number of encounters.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Schnipper, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Jeffrey L Schnipper, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No specimens will be collected for this study and no identifiable data will be shared with research collaborators outside Partners. Data collected through this study may be used to further research in post-operative opioid use, but all data will be de-identified prior to storage and use by collaborators.